CLINICAL TRIAL: NCT02374476
Title: Bipolar Catheter Ablation for the Treatment of Refractory Scar-Related Ventricular Arrhythmia
Brief Title: Bipolar Ventricular Tachycardia (VT) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Srinivas Dukkipati (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Srinivas Dukkipati, Co-Director EP Service, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 14-1827
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Results first posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Ventricular Tachycardia
Keywords: VT; Refractory VT; VT Storm; Ventricular Fibrillation; V Fib; VF
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Bipolar Ablation (Experimental): All patients who meet inclusion criteria and have VT not terminable with unipolar ablation will undergo bipolar ablation.
  Interventions: Device: Bipolar Ablation
- Registry (Active Comparator): Participants in Patient Registry after standard radiofrequency (VT) unipolar radiofrequency (RF) ablation was successful
  Interventions: Device: Bipolar Ablation

INTERVENTIONS:
Device: Bipolar Ablation — Patients will undergo bipolar ablation if unipolar ablation unsuccessful

SUMMARY:
This non-randomized study will examine the safety and efficacy of irrigated bipolar radiofrequency (RF) ablation in the treatment of ventricular tachycardia (VT) in patients for whom standard VT unipolar RF ablation has been unsuccessful. VT is a serious abnormality of the heart's electrical system. Ablation is a procedure that cauterizes heart tissue using catheters (long tubes that can be moved within or along the outside of the heart). Cauterizing the heart tissue is accomplished by using heat to damage the abnormal heart tissue that is not working well so that it can stop affecting the rest of the heart. Usually, heat is delivered using a unipolar catheter, in which energy travels from the catheter tip to a grounding pad. This research study seeks to find out if a bipolar ablation catheter, in which the energy travels between two catheter tips on either side of the heart muscle, can be used to eliminate the arrhythmia when the unipolar ablation is unsuccessful. The hypothesis is that the increased current density and improved rates of transmural lesion creation seen with bipolar RF ablation will lead to successful arrhythmia termination with minimal or no increased risk of complication.

DETAILED DESCRIPTION:
STUDY OBJECTIVE This study will examine the role of irrigated bipolar radiofrequency (RF) ablation for the treatment of intramural ventricular tachycardia in patients who have failed standard unipolar RF ablation. The hypothesis is that the increased current density and improved rates of transmural lesion creation seen with bipolar RF ablation will lead to successful arrhythmia termination with minimal or no increased risk of complication.

INTRODUCTION, RATIONALE Radiofrequency (RF) ablation is the most commonly employed method for the catheter treatment of cardiac arrhythmias. Myocardial scar serves as the most frequent substrate for the genesis of both atrial and ventricular arrhythmia. Such scar frequently contains surviving myocyte bundles interspersed with fibrotic tissue, which leads to slow conduction. Areas of denser fibrosis cause conduction block. When appropriately arranged, conduction through or around these scars leads to the creation of a "reentry" circuit through which an arrhythmia is generated and maintained. Each reentry circuit contains within it an area called the isthmus, a portion of the circuit located in a position intimately related to the scar border zone. Electrical activation travels slowly through the isthmus before breaking out into normal myocardium. Ablation at the site of an isthmus will terminate a reentrant tachycardia.

A variety of techniques, including electroanatomic mapping and activation, entrainment, and substrate mapping, are employed during electrophysiologic (EP) study to identify areas of myocardial scar and potential isthmus sites. Points or lines of ablation using RF energy are then created in an attempt to interrupt the reentry circuit. Typically, unipolar RF energy is applied via a catheter tip electrode to the endocardial or epicardial surface of the heart and grounded via an electrode pad placed on the patient's skin. RF energy in this setting is dispersed through the entirety of the tissue between catheter tip and grounding pad. The standard 7-French, 4-mm tip catheters are highly successful at ablating circuits located within a few millimeters of the catheter tip. A focal, 1mm area of resistive heating occurs within the myocardium immediately in contact with the catheter tip; myocardial cell death occurs several millimeters more deeply through passive, conductive heating, which spreads outward from the contact point.

While the standard catheter is effective at the ablation of superficial arrhythmias, it has proven more problematic when used for deep myocardial sites or for creating transmural lesions. A number of alternatives have been developed in an attempt to access these sites. 8-mm or 10-mm catheter tips are able to create larger zones of resistive heating, delivering direct RF energy to a larger area of myocardium. A larger interface between catheter tip and blood improves cooling and allows for the delivery of more power without a rise in impedence. The clinical use of these larger catheters can, however, be limited by rapid temperature rises at the catheter-tissue interface, resulting in thrombus formation, char, and "steam pop" rupture of the endocardial surface. The use of irrigated ablation catheters have improved upon the ability to deliver RF energy without a sustained rise in impedance. Both open irrigated- and closed-loop irrigated catheters circulate saline along the catheter tip-myocardial interface, allowing for continued delivery of RF current without thrombus formation at the endocardial surface. Intramyocardial temperature rises accordingly without a concomitant endocardial temperature surge, creating larger and deeper myocardial ablation zones. Catheters featuring a retractable needle tipped electrode with intramyocardial saline infusion have also shown promise as a means of accessing deep myocardial circuits in ventricular tachycardia ablation, but are not currently available in the US. Transcoronary ethanol ablation has also been employed with moderate success in patients with arrhythmias resistant to endocardial catheter ablation. This technology, however, grants only limited control over the size of the resulting infarct and is restricted by the need for perfusion of the scar zone by an accessible coronary artery.

Nevertheless, there remain occasions in which an arrhythmia cannot be eliminated by standard unipolar ablation technique. This is seen most frequently due to deep intramural ventricular tachycardia, sometimes encountered following myocardial infarction. Both standard and alternative ablation strategies are frequently either unavailable or inadequate for termination of these arrhythmias.

Recently, several centers have employed irrigated bipolar ablation (BA) to target arrhythmias not amenable to unipolar ablation. During BA, two catheters are connected to either pole of an RF generator, allowing either catheter to function as the "active" catheter and the other the "return" catheter. Rather than being dispersed between the catheter tip and a distant grounding pad, BA concentrates energy between two catheter tips positioned on opposing sides of a target scar. BA may thus improve lesion transmurality through synergistic, simultaneous heating and increased current density leading to concentrated thermal injury.

Initial experience in the use of BA technology in mammalian hearts demonstrated that it could successfully be applied to create discrete areas of myocardial necrosis with minimal risk of complication. When compared to unipolar ablation, several studies suggested that BA could create larger areas of necrosis and transmural lesions with only rare episodes of perforation. Subsequent experience in human hearts was predominantly surgical: a large number of observational studies and reviews demonstrated the effectiveness and safety of BA in patients undergoing pulmonary vein isolation and Cox-Maze surgery as either isolated procedures or as adjuncts to valve replacement or coronary artery bypass surgery.

Despite its broad use during surgical ablation, the application of BA during catheter-based therapies is limited. Recently, our group demonstrated the utility of BA in both an in vitro model and in a series of patients with arrhythmia resistant to unipolar ablation. When compared to unipolar RF ablation, BA was found to be more likely to achieve transmural lesions in a porcine heart model (33% vs 82%, respectively, p = 0.001) and could do so in tissue up to 25 mm thickness. Clinically, all septal atrial flutters, 5 of 6 septal VTs, and 2 of 4 free-wall VTs were successfully acutely terminated.

The proposed study will further examine the role of BA in patients with ventricular tachycardia resistant to standard ablation techniques.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* The study will include all forms of scar VT--both ischemic (post-myocardial infarction) and non-ischemic (eg sarcoid, amyloid, dilated)--as determined by cardiac MRI and/or voltage mapping at the time of VT ablation.
* Intramural VT not terminable with unipolar ablation once enrolled in the Bipolar study or previous failed unipolar ablation within 6 months prior to enrollment.
* Ability to understand the requirements of the study and sign the informed consent form.
* Willingness to adhere to study restrictions and comply with all post- procedural follow-up requirements
* Projected lifespan greater than 1 year.

Exclusion Criteria:

* Tissue Thickness less than 5 mm as assessed by electroanatomic mapping, CT, or MRI.
* MI or CABG within 6 weeks.
* NYHA Class IV CHF.
* Women known to be pregnant or to have positive beta-HCG.
* Participation in another study that would interfere with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2015-02-18 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Dukkipati, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (6):
- United States (6):
  - Loyola University Medical Center, Maywood, Illinois
  - Brigham & Womans Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: All patients who met inclusion criteria and have VT not terminable with unipolar ablation underwent bipolar ablation.
- Bipolar Ablation: Participants who underwent bipolar ablation after unipolar ablation unsuccessful
Period: VT Induced Ablation
Arm/Group | All Patients | Bipolar Ablation | Registry
Started | 145 | 0 | 0
Completed | 109 | 0 | 0
Not Completed | 36 | 0 | 0
Not completed — Screening Failures | 36 | 0 | 0
Period: Arm Assignment
Arm/Group | All Patients | Bipolar Ablation | Registry
Started | 0 | 49 | 60
Completed | 0 | 49 | 59
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Patient Registry: Participants in Patient Registry after standard radiofrequency (VT) unipolar radiofrequency (RF) ablation was successful
- Total: Total of all reporting groups
Arm/Group | Bipolar Ablation | Patient Registry | Total
Number analyzed (Participants) | 49 | 60 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.88 (11.29) | 63.1 (11.31) | 63 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 47 | 54 | 101
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Freedom From Recurrent Ventricular Tachycardia (VT)
Description: Freedom from recurrent VT at 6 months, defined as sustained ventricular tachycardia lasting longer than 30 seconds and identified due to clinical symptoms or during device interrogation.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bipolar Ablation | Patient Registry
Number analyzed (Participants) | 49 | 60
Participants | 16 | 29

2. Secondary Outcome: Number of Procedural Complications
Description: Total number of procedural complications which includes death, stroke, MI, heart failure, conduction abnormalities, pericardial effusion requiring drainage, hematoma, pseudoaneurysm
Time Frame: 6 months
Measure: Number; unit: events
Arm/Group | Bipolar Ablation | Patient Registry
Number analyzed (Participants) | 49 | 60
events | 31 | 19

3. Secondary Outcome: Number of Participants With Post-ablation Inducibility of VT
Description: Number of participants to indicate incidence of the induction of any sustained arrhythmia post-ablation, with a duration > 15 seconds of monomorphic VT (MMVT). Post ablation inducibility is measured via program stimulation.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bipolar Ablation | Patient Registry
Number analyzed (Participants) | 49 | 60
Participants | 6 | 5

4. Secondary Outcome: Time to Arrhythmia Termination for the Bipolar Group Only
Description: When bipolar ablation is performed during ongoing Ventricular Tachycardia (VT), the time to termination is the amount of ablation time that was necessary to cause VT to stop (terminate)
Time Frame: through termination, up to 60 seconds
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Bipolar Ablation: Bipolar Ablation: Patients underwent bipolar ablation when unipolar ablation unsuccessful
Arm/Group | Bipolar Ablation
Number analyzed (Participants) | 49
seconds | 14.33 (10.29)

5. Secondary Outcome: Total Duration of Bipolar Ablation
Description: Duration of bipolar ablation is the total procedure time
Time Frame: average of 345 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Bipolar Ablation | Patient Registry
Number analyzed (Participants) | 49 | 60
minutes | 342.22 (133.82) | 317.33 (128.98)

6. Secondary Outcome: Number of of Participants With Mortality
Description: Number of participant from all cause mortality
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bipolar Ablation | Patient Registry
Number analyzed (Participants) | 49 | 60
Participants | 9 | 5

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Bipolar Ablation | Patient Registry
All-Cause Mortality (participants affected / at risk) | 9/49 | 5/60
Serious Adverse Events (participants affected / at risk) | 26/49 | 25/60
Other Adverse Events (participants affected / at risk) | 14/49 | 8/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bipolar Ablation (N=49) | Patient Registry (N=60)
Cardiac Tamponade (Cardiac disorders) | 4 | 0
Recurrent Ventricular Tachycardia (Cardiac disorders) | 9 | 10
Pulmonary Embolism Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pericardial Effusion due to myocardial performation (Cardiac disorders) | 1 | 0
Left Ventricular Thrombus (Cardiac disorders) | 1 | 1
Pericardial Effusion (Cardiac disorders) | 6 | 1
Hemorrhagic Shock (Cardiac disorders) | 2 | 0
New Incessant Ventricular Tachycardia (Cardiac disorders) | 2 | 0
Pericarditis (Cardiac disorders) | 2 | 0
Hemothorax (Cardiac disorders) | 1 | 0
Cardiac Arrest/anoxic brain injury (Cardiac disorders) | 1 | 0
Implantable Cardioverter Defibrillator Shock (Cardiac disorders) | 1 | 0
Chest pain/Fever (General disorders) | 2 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lower Extremity Swelling/Weight Gain (General disorders) | 1 | 0
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 2 | 0
Hemodynamic decompensation/cardiac arrest post procedure (Cardiac disorders) | 1 | 0
Total Artificial Heart Implantation/Severe atherosclerotic Coronary Artery Disease (Cardiac disorders) | 1 | 0
Acute MI (Cardiac disorders) | 1 | 0
Recurrent Ventricular Tachycardia/LVAD Implantation (Cardiac disorders) | 1 | 0
Aortic Regurgitation requiring valve replacement (Cardiac disorders) | 1 | 0
Generator change (Cardiac disorders) | 2 | 0
Lead revision due to increased defibrillation threhold (Cardiac disorders) | 1 | 0
Heart Transplant (Cardiac disorders) | 1 | 0
Hemoperitoneum (Vascular disorders) | 2 | 0
Cardiogenic Shock/Septic Shock (Cardiac disorders) | 1 | 0
Gastrointestinal Bleed/Melena (Gastrointestinal disorders) | 1 | 0
Pulseless Electrical Activity (Cardiac disorders) | 1 | 0
Oopharyngeal swallow dysfunction (General disorders) | 1 | 0
Hypercarbia and Fluid Overload (Cardiac disorders) | 1 | 0
Congestive Heart Failure (Cardiac disorders) | 1 | 3
Right Femoral Artery Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Fluid Overload (Cardiac disorders) | 1 | 1
Right Ventricular Failure (Cardiac disorders) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Hypoxic Brain Injury (Nervous system disorders) | 1 | 0
recurrent ventricular tachycardia with biventricular failure (Cardiac disorders) | 0 | 1
renal failure (Renal and urinary disorders) | 0 | 1
new incessant ventricular tachycardia with redo ablation (Cardiac disorders) | 0 | 1
back pain/diaphoresis/hematuria (General disorders) | 0 | 1
pre-syncope and elevated cardiact enzymes (Cardiac disorders) | 0 | 1
recurrent ventricular tachycardia/end stage heart failure (Cardiac disorders) | 0 | 1
pneumoperitoneum, renal failure (intolerable to dialysis) (Renal and urinary disorders) | 0 | 1
congestive heart failure/fluid overload (Cardiac disorders) | 0 | 1
cerebrovascular accident/encephalopahty (Nervous system disorders) | 0 | 1
orchitis (Infections and infestations) | 0 | 1
food poisoining (General disorders) | 0 | 1
cardiogenic shock (Cardiac disorders) | 0 | 1
left femoral pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
slurred speech (Nervous system disorders) | 0 | 1
right subclavian/axillary thrombosis (Vascular disorders) | 0 | 1
oropharynx bleeding (Injury, poisoning and procedural complications) | 0 | 1
hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
gastrointestinal bleed (Gastrointestinal disorders) | 0 | 1
hemo-pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
lead modification (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bipolar Ablation (N=49) | Patient Registry (N=60)
Complete Heart Block (Cardiac disorders) | 6 | 2
Acute Kidney Injury (Renal and urinary disorders) | 2 | 3
Volume Overload (Cardiac disorders) | 3 | 2
Groin Hematoma (Vascular disorders) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Post Ablation Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT02374476/Prot_SAP_000.pdf